CLINICAL TRIAL: NCT04457024
Title: Tennis Elbow Patients Undergoing Closed Therapy Can Easily Cause Tendon Tear
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019143
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Tennis Elbow; MRI; Hyperlipidemia
MeSH Terms: conditions — Tennis Elbow; Hyperlipidemias | interventions — Statistics as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: classification statistics — Without any intervention

SUMMARY:
To explore whether there is a difference in the rate of tendon tear after hyperlipemia in tennis elbow patients and those with normal blood lipids after closed treatment, which provides clues for further exploration of its mechanism. 1. Collect data from 108 cases of tennis elbow patients treated at the Institute of Sports Medicine, Peking University Third Hospital from January 2010 to December 2018 at the Institute of Sports Medicine, Peking University Third Hospital. Statistics included the sex, age, BMI, number of closures, total cholesterol, triglycerides, low-density lipoprotein, high-density lipoprotein. 2. Retrieve the MRI imaging data of the above-mentioned patients, and use the extensor tendon at the humerus to see if there is a tear as an observation indicator. Analyze the difference of tendon tear after closed treatment in patients with high blood fat and normal blood fat.

ELIGIBILITY:
Inclusion Criteria:

* All patients with tennis elbows in our hospital

Exclusion Criteria:

* none

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: In order to rule out the influence of the imbalance between height and weight on blood lipids, the difference between the case group and the control group was analyzed after adjusting the height and weight covariates using the Generalized Linear Model.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Use MRI to assess whether the tendon is torn | 3 months
  One sports medicine surgeon and one musculoskeletal radiologists, being blinded to the patients' information, reviewed the elbow MRI independently. The common extensor tendon (CET) abnormalities were evaluated on axial and coronal fat-suppressed T2-weighted FSE image. Tendinosis group was defined as an increased signal intensity, but lower than the fluid signal on T2-weighted images and/ or an increased tendon thickness. Tendon tear group contain a partial thickness tear defined as a region with fluid-signal-intensity that extended partway across the tendon and a full thickness tear appeared as a gap of fluid-signal-intensity across the entire tendon substance.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Univerisity Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No